CLINICAL TRIAL: NCT02981407
Title: Myocardial Ischemia and Transfusion
Acronym: MINT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Pittsburgh (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Principal Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro20160000722; 1U01HL133817-01 (NIH)
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Myocardial Infarction; Anemia
Keywords: Red Blood Cell Transfusion; Anemia; Heart Disease; Cardiovascular Disease
MeSH Terms: conditions — Myocardial Infarction; Anemia; Heart Diseases; Cardiovascular Diseases | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liberal Transfusion Strategy (Active Comparator): Red blood cell transfusion - One unit of packed red cells is transfused following randomization followed by enough red blood cell units to raise the hemoglobin concentration above 10 g/dL any time the hemoglobin concentration is detected to be below 10g/dL during the hospitalization for up to 30 days.
  Interventions: Biological: Red Blood Cell Transfusion
- Restrictive Transfusion Strategy (Active Comparator): Permitted to receive a red blood cell transfusion if the blood count is below 8 g/dL and the physician believes it is in the patient's best interest. A transfusion will be strongly recommended if the blood count drops to less than 7 g/dL. If the patient has symptoms of angina (e.g., chest discomfort described as pressure or heaviness) that do not go away with medication, a blood transfusion will be ordered regardless of the blood count.
  Interventions: Biological: Red Blood Cell Transfusion

INTERVENTIONS:
Biological: Red Blood Cell Transfusion — Transfusion of packed red blood cell units

SUMMARY:
The purpose of this study is to compare two red blood cell transfusion strategies (liberal and restrictive) for patients who have had an acute myocardial infarction and are anemic.

DETAILED DESCRIPTION:
In most clinical settings, evidence suggests it is safe to wait to give a blood transfusion. However, for those who have suffered a heart attack, there is a lack of high quality evidence to guide transfusions. This 3500 subject multi-center randomized trial will fill that void.

Hospital inpatients diagnosed with myocardial infarction who have blood counts less than 10 g/dL are randomized to receive either a liberal or a restrictive transfusion strategy.

Patients randomized to the liberal transfusion strategy will receive a red blood cell transfusion anytime there is a blood count of less than 10 g/dL.

Patients randomized to the restrictive transfusion strategy are permitted to receive a blood transfusion if the blood count is below 8 g/dL and the physician believes it is in the patient's best interest. A transfusion will be strongly recommended if the blood count drops to less than 7 g/dL. If the patient has symptoms of angina (e.g., chest discomfort described as pressure or heaviness) that do not go away with medication, a blood transfusion is ordered regardless of the blood count.

The transfusions strategies will be maintained until hospital discharge for a maximum of 30 days.

Patients will be followed for 30 days for clinically relevant outcomes. Vital status will be confirmed at 180 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Either ST segment elevation myocardial infarction or Non ST segment elevation myocardial infarction consistent with the 3rd Universal Definition of Myocardial Infarction criteria that occurs on admission or during the index hospitalization
* Hemoglobin concentration less than 10 g/dL at the time of random allocation
* Patient physician believes that both of the transfusion strategies are consistent with good medical care for the patient

Exclusion Criteria:

* Uncontrolled acute bleeding at the time of randomization defined as the need for uncrossed or non-type specific blood
* Decline blood transfusion
* Scheduled for cardiac surgery during the current admission
* Receiving only palliative treatment
* Known that follow-up will not be possible at 30 days
* Previously participated in MINT
* Currently enrolled in a competing study that interferes with the intervention or follow-up of MINT or enrolled in a competing study that has not been approved by the local Institutional Review Board
* Patient physician does not believe the patient is an appropriate candidate for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3506 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School; Maria Mori Brooks, PhD, Principal Investigator — University of Pittsburgh
Locations (133):
- United States (60):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas Medical Sciences (UAMS) Hospital, Little Rock, Arkansas
  - VAGLAHS, Los Angeles, California
  - Danbury Hospital, Danbury, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - AMITA Health, Hinsdale, Illinois
  - Saint Luke's Mid America Heart, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Health System, Ypsilanti, Michigan
  - Essentia Health, Duluth, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Minneapolis Heart Institute (Foundation), Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Washington University, St Louis, Missouri
  - Copper University Hospital, Camden, New Jersey
  - Hackensacjk University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical, Neptune City, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Southside Hospital, Bay Shore, New York
  - NYP Brooklyn Methodist, Brooklyn, New York
  - New York Presbyterian/Queens, Flushing, New York
  - Westchester Medical Center, Hawthorne, New York
  - North Shore University Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - NYU Langone Medical Center, Bellevue Hospital, New York, New York
  - Lenox Hilll Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Northwell Staten Island Hopsital, Staten Island, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Durham Va, Durham, North Carolina
  - WakeMed Health and Hospital, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - PENN Presbyterian Medical Cente, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Greenville Health System, Greenville, South Carolina
  - The Memphis VAMC, Memphis, Tennessee
  - Baylor St Luke's Medical Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (4):
  - Flinders Medical Centre, Bedford Park
  - Concord Repatriation General Hospital, Concord
  - Gosford Hospital, Gosford
  - Royal Perth Hospital, Perth
- Brazil (18):
  - Instituto de Ensino e Pesquisa do Hospital da Bahia, Pituba, Salvador
  - Hospital de Base de Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Felício Rocho, Belo Horizonte
  - Instituto Orizonti, Belo Horizonte
  - Instituto de Ensino e Pesquisa do Hospital do Coração do Brasil, Brasília
  - Hospital Vera Cruz, Campinas
  - Santa Casa de Marília, Cascata
  - Sociedade Hospitalar Angelina Caron, Centro
  - Hospital Maternidade e Pronto Socorro Santa Lúcia, Poços de Caldas
  - Instituto de Cardiologia do RS, Porto Alegre
  - Hospital Agamenon Magalhães, Recife
  - Pronto Socorro Cardiológico de Pernambuco Prof. Luiz Tavares- PROCAPE, Recife
  - Hospital Cárdio Pulmonar, Salvador
  - Hospital Universitário Professor Edgard Santos, Salvador
  - Hospital de Base de Rio Preto, São José do Rio Preto
  - Hospital São Paulo, São Paulo
  - Hospital de Clínicas da UFTM, Uberaba
  - Hospital das Clinicas da UFU, Uberlândia
- Canada (27):
  - Foothills Medical Centre, Calgary, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QE II Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Hamilton St. Joseph's Health, Hamilton, Ontario
  - St. Joseph's Health Centre, Hamilton, Ontario
  - University Hospital - LHSC, London, Ontario
  - Victoria Hospital - LHSC, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Victoria Heart Institute, Victoria, Ontario
  - Hôpital Charles Lemoyne, Greenfield Park, Quebec
  - Hotel-Dieu de Levis, Lévis, Quebec
  - Centre Hosp. Universitaire de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Quebec Heart and Lung Institute, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - General Hospital Trois-Rivièrs, Trois-Rivières, Quebec
  - Regina General Hospital, Regina, Saskatchewan
- France (18):
  - CHRU Tours -Hôpital Trousseau, Chambray-lès-Tours
  - CH Chartres - Chartres, Chartres
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU le Bocage - Dijon, Dijon
  - La Tronche Hôpital Michallon, La Tronche
  - Centre Hospitalier Universitaire de Lille, Lille
  - CHU Arnaud de Villeneuve - Montpellier, Montpellier
  - CHU Nancy, Nancy
  - Hôpital Pasteur, Nice
  - Hôpital Universitaire Carémeau (CHU Carémeau), Nîmes
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital BICHAT- APHP, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Haut Lévêque, Pessac
  - CHU Poitiers - Poitiers, Poitiers
  - Hôpital Charles Nicolle- Rouen, Rouen
  - Hôpital Rangueil, Toulouse
- New Zealand (6):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Gisborne Hospital, Gisborne
  - Nelson Hospital, Nelson
  - Taranaki Hospital, New Plymouth
  - Whangarei Hospital, Whangarei

IPD SHARING:
Plan to Share IPD: Yes
Limited access data (i.e., records without personal identifiers) will be prepared by the Data Coordinating Center (DCC) and sent to the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) within 3 years after the end of the final patient follow-up or 2 years after the main paper of the trial has been published, whichever comes first. The Trial data set will include baseline patient characteristics, follow-up status, and clinical outcome data. The data will be released to requesting institutions and investigators in accordance with BioLINCC policy.

REFERENCES:
- [Background] Carson JL, Brooks MM, Abbott JD, Chaitman B, Kelsey SF, Triulzi DJ, Srinivas V, Menegus MA, Marroquin OC, Rao SV, Noveck H, Passano E, Hardison RM, Smitherman T, Vagaonescu T, Wimmer NJ, Williams DO. Liberal versus restrictive transfusion thresholds for patients with symptomatic coronary artery disease. Am Heart J. 2013 Jun;165(6):964-971.e1. doi: 10.1016/j.ahj.2013.03.001. Epub 2013 Apr 8. PMID 23708168
- [Background] Carson JL, Guyatt G, Heddle NM, Grossman BJ, Cohn CS, Fung MK, Gernsheimer T, Holcomb JB, Kaplan LJ, Katz LM, Peterson N, Ramsey G, Rao SV, Roback JD, Shander A, Tobian AA. Clinical Practice Guidelines From the AABB: Red Blood Cell Transfusion Thresholds and Storage. JAMA. 2016 Nov 15;316(19):2025-2035. doi: 10.1001/jama.2016.9185. PMID 27732721
- [Background] Carson JL, Brooks MM, Chaitman BR, Alexander JH, Goodman SG, Bertolet M, Abbott JD, Cooper HA, Rao SV, Triulzi DJ, Fergusson DA, Kostis WJ, Noveck H, Simon T, Steg PG, DeFilippis AP, Goldsweig AM, Lopes RD, White H, Alsweiler C, Morton E, Hebert PC; MINT Investigators. Rationale and design for the myocardial ischemia and transfusion (MINT) randomized clinical trial. Am Heart J. 2023 Mar;257:120-129. doi: 10.1016/j.ahj.2022.11.015. Epub 2022 Nov 20. PMID 36417955
- [Background] Carson JL, Brooks MM, Hebert PC, Goodman SG, Bertolet M, Glynn SA, Chaitman BR, Simon T, Lopes RD, Goldsweig AM, DeFilippis AP, Abbott JD, Potter BJ, Carrier FM, Rao SV, Cooper HA, Ghafghazi S, Fergusson DA, Kostis WJ, Noveck H, Kim S, Tessalee M, Ducrocq G, de Barros E Silva PGM, Triulzi DJ, Alsweiler C, Menegus MA, Neary JD, Uhl L, Strom JB, Fordyce CB, Ferrari E, Silvain J, Wood FO, Daneault B, Polonsky TS, Senaratne M, Puymirat E, Bouleti C, Lattuca B, White HD, Kelsey SF, Steg PG, Alexander JH; MINT Investigators. Restrictive or Liberal Transfusion Strategy in Myocardial Infarction and Anemia. N Engl J Med. 2023 Dec 28;389(26):2446-2456. doi: 10.1056/NEJMoa2307983. Epub 2023 Nov 11. PMID 37952133
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Prochaska MT, Portela GT, Brooks MM, Fergusson DA, Hebert PC, Polonsky TS, Caixeta A, Cooper HA, Crozier I, Daneault B, Kim S, Bainey KR, de Barros E Silva P, Goldfarb M, Gupta R, Rao SV, Fonteles Ritt LE, Simon T, Carson JL. Transfusion Strategy Effect on Quality of Life in Patients With Myocardial Infarction and Anemia: A Secondary Analysis of the MINT Randomized Clinical Trial. JAMA Intern Med. 2025 Aug 1;185(8):947-954. doi: 10.1001/jamainternmed.2025.0654. PMID 40459491
- [Derived] Rao SV, Brooks MM, D'Agostino HEA, Steg PG, Simon T, Aronow HD, Goldsweig AM, Malik S, Alsweiler C, Ho KKL, Dehghani P, Caixeta A, Quraishi AR, Robinson S, Traverse JH, Siddiqi O, Fergusson DA, Potter BJ, Schulman-Marcus J, Keating FK, Carson JL; MINT Trial Investigators. Effect of Red Blood Cell Transfusion Strategy on Clinical Outcomes Among Patients With Acute Myocardial Infarction Undergoing Revascularization: A Prespecified Analysis of the MINT Trial. Circ Cardiovasc Interv. 2025 May;18(5):e015249. doi: 10.1161/CIRCINTERVENTIONS.125.015249. Epub 2025 Mar 30. PMID 40159118
- [Derived] Goldsweig AM, Kostis WJ, Herbert BM, Bouleti C, Potter BJ, Strom JB, Benatar J, Huynh T, Vallurupalli S, Figueiredo EL, Abbott JD, Cooper HA, DeFilippis AP, Fergusson DA, Goodman SG, Hebert PC, Lopes RD, Rao SV, Simon T, Carson JL, Brooks MM, Alexander JH; MINT Investigators. Blood Transfusion in Patients With Acute Myocardial Infarction, Anemia, and Heart Failure: Lessons From MINT. Circ Heart Fail. 2025 Apr;18(4):e012495. doi: 10.1161/CIRCHEARTFAILURE.124.012495. Epub 2025 Mar 26. PMID 40135329
- [Derived] Portela GT, Ducrocq G, Bertolet M, Alexander JH, Goodman SG, Glynn S, Strom JB, Swanson SA, Lemesle G, Rao SV, Tessalee M, Polonsky TS, Goldfarb M, Traverse JH, Uhl L, Herbert BM, Silvain J, Carson JL, Brooks MM; MINT Trial Investigators. Individualized transfusion decisions to minimize adverse cardiovascular outcomes in patients with acute myocardial infarction and anemia. Am Heart J. 2025 Apr;282:146-155. doi: 10.1016/j.ahj.2025.01.009. Epub 2025 Jan 17. PMID 39826701
- [Derived] Strom JB, Herbert BM, Bertolet M, Brooks MM, Malik SA, Lemesle G, Madan M, Steg PG, Hebert PC, Traverse JH, White HD, Alsweiler C, Gupta R, Ritt LEF, Menegus MA, Alexander JH, Lopes RD, Chaitman BR, Carson JL; MINT Trial Investigators. Restrictive or Liberal Blood Transfusion in Patients with Myocardial Infarction and CKD. J Am Soc Nephrol. 2025 Jun 1;36(6):1116-1125. doi: 10.1681/ASN.0000000595. Epub 2025 Jan 9. PMID 39786901
- [Derived] Carrier FM, Cooper HA, Portela GT, Bertolet M, Lemesle G, Prochaska M, Kim S, Alexander JH, Crozier I, Ducrocq G, Quadros AS, Bagai A, Dracoulakis M, Madan M, Brooks MM, Carson JL, Hebert PC; MINT Investigators. Anemia Acuity Effect on Transfusion Strategies in Acute Myocardial Infarction: A Secondary Analysis of the MINT Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2442361. doi: 10.1001/jamanetworkopen.2024.42361. PMID 39485351
- [Derived] Portela GT, Carson JL, Swanson SA, Alexander JH, Hebert PC, Goodman SG, Steg PG, Bertolet M, Strom JB, Fergusson DA, Simon T, White HD, Cooper HA, Abbott JD, Rao SV, Chaitman BR, Fordyce CB, Lopes RD, Daneault B, Brooks MM; MINT Investigators. Effect of Four Hemoglobin Transfusion Threshold Strategies in Patients With Acute Myocardial Infarction and Anemia : A Target Trial Emulation Using MINT Trial Data. Ann Intern Med. 2024 Nov;177(11):1489-1498. doi: 10.7326/M24-0571. Epub 2024 Oct 1. PMID 39348705
- [Derived] Simon T, Herbert BM, Brooks MM, Goodman SG, Alexander JH, Steg PG, Lopes RD, Ghafghazi S, Bouleti C, Cooper HA, McCamant EL, Bainey KR, Aronow HD, Abbott JD, Alsweiler C, Bertolet M, Fergusson DA, Goldsweig AM, Hebert PC, Carson JL; MINT Trial Investigators. Restrictive or Liberal Transfusion Strategy in Patients With Acute Myocardial Infarction and Anemia: 6-Month Mortality in the MINT Trial. Circulation. 2024 Sep 24;150(13):1064-1066. doi: 10.1161/CIRCULATIONAHA.124.069917. Epub 2024 Sep 2. No abstract available. PMID 39221566
- [Derived] DeFilippis AP, Abbott JD, Herbert BM, Bertolet MH, Chaitman BR, White HD, Goldsweig AM, Polonsky TS, Gupta R, Alsweiler C, Silvain J, de Barros E Silva PGM, Hillis GS, Daneault B, Tessalee M, Menegus MA, Rao SV, Lopes RD, Hebert PC, Alexander JH, Brooks MM, Carson JL, Goodman SG; MINT Investigators. Restrictive Versus Liberal Transfusion in Patients With Type 1 or Type 2 Myocardial Infarction: A Prespecified Analysis of the MINT Trial. Circulation. 2024 Dec 3;150(23):1826-1836. doi: 10.1161/CIRCULATIONAHA.124.071208. Epub 2024 Aug 29. PMID 39206549
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Started | 1757 | 1749
Data at 30 Days Post Randomization | 1755 (37 of these participants had incomplete data for some outcomes) | 1749 (20 of these participants had incomplete data for some outcomes)
Completed | 1755 | 1749
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy | Total
Number analyzed (Participants) | 1755 | 1749 | 3504
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (11.6) | 72.2 (11.5) | 72.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 819 | 774 | 1593
  Male | 936 | 975 | 1911
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 134 | 119 | 253
  Not Hispanic or Latino | 1434 | 1445 | 2879
  Unknown or Not Reported | 187 | 185 | 372
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1245 | 1229 | 2474
  Black | 223 | 217 | 440
  Other | 115 | 129 | 244
  Unknown | 172 | 174 | 346
Type of Myocardial Infarction [Count of Participants; unit: Participants] — Type 1 myocardial infarction occurs in those with atherosclerotic plaque rupture and thrombosis. Type 2 myocardial infarction occurs due to myocardial oxygen supply and demand imbalance. Other includes myocardial infarction due to stent thrombosis or restenosis.
  Participants
    Type 1 | 730 | 730 | 1460
    Type 2 | 988 | 967 | 1955
    Other or Unknown | 37 | 52 | 89
ST or Non-ST-Elevation Myocardial Infarction [Count of Participants; unit: Participants]
  STEMI | 337 | 319 | 656
  NSTEMI | 1418 | 1430 | 2848
History of Myocardial Infarction [Count of Participants; unit: Participants]
  Yes | 549 | 589 | 1138
  No | 1206 | 1160 | 2366
History of Percuatneous Coronary Intervention [Count of Participants; unit: Participants]
  Yes | 577 | 623 | 1200
  No | 1177 | 1126 | 2303
  Unknown | 1 | 0 | 1
History of Coronary Artery Bypass Surgery [Count of Participants; unit: Participants]
  Yes | 390 | 372 | 762
  No | 1365 | 1377 | 2742
History of Heart Failure [Count of Participants; unit: Participants]
  Yes | 539 | 527 | 1066
  No | 1216 | 1222 | 2438

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Mortality or Nonfatal Myocardial Reinfarction
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 255 | 295

2. Secondary Outcome: All-cause Mortality
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 146 | 173

3. Secondary Outcome: Myocardial Reinfarction
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 126 | 149

4. Secondary Outcome: Composite of All-cause Mortality, Nonfatal Myocardial Reinfarction, Ischemia Driven Unscheduled Coronary Revascularization, or Readmission to the Hospital for Ischemic Cardiac Diagnosis
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 305 | 342

5. Other Pre Specified Outcome: Composite of All-cause Mortality,Nonfatal Myocardial Reinfarction, or Unstable Angina
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 300 | 338

6. Other Pre Specified Outcome: Ischemia Driven Unscheduled Coronary Revascularization
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 39 | 43

7. Other Pre Specified Outcome: Unscheduled Readmission to Hospital for Ischemic Cardiac Diagnosis
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Heart Failure
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 111 | 102

9. Other Pre Specified Outcome: Unscheduled Readmission to Hospital for Any Reason
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Stroke
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 26 | 30

11. Other Pre Specified Outcome: Pulmonary Embolism or Deep Venous Thrombosis
Time Frame: Within 30 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
Number analyzed (Participants) | 1755 | 1749
Participants | 34 | 26

12. Other Pre Specified Outcome: Bleed
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pneumonia
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Blood Stream Infection
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Urinary Tract Infection
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Length of Hospital Stay Post Randomization
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Number of Days Post Randomization in Intensive Care Unit
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Patient Reported Quality of Life
Description: EuroQol questionnaire
Time Frame: Within 30 days of randomization
Reporting Status: Not Posted

19. Other Pre Specified Outcome: All-cause Mortality
Time Frame: Within 6 months of randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through 30 days and death was collected through 180 days
Description: Research staff contacted participants/proxies at 30 days to collect clinical events and at 180 days to determine vital status
Arm/Group | Liberal Transfusion Strategy | Restrictive Transfusion Strategy
All-Cause Mortality (participants affected / at risk) | 353/1755 | 376/1749
Serious Adverse Events (participants affected / at risk) | 699/1755 | 723/1749
Other Adverse Events (participants affected / at risk) | 330/1755 | 348/1749
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal Transfusion Strategy (N=1755) | Restrictive Transfusion Strategy (N=1749)
Myocardial Infarction (Cardiac disorders) | 126 (126) | 149 (149)
Heart Failure (Cardiac disorders) | 111 (111) | 102 (102)
Super ventricular tachycardia (Cardiac disorders) | 28 (28) | 27 (27)
Ventricular tachycardia (Cardiac disorders) | 56 (56) | 59 (59)
Ventricular fibrillation (Cardiac disorders) | 14 (14) | 19 (19)
Cardiac arrest (Cardiac disorders) | 45 (45) | 69 (69)
Mobitz type 2 atrial ventricular block (Cardiac disorders) | 13 (13) | 15 (15)
Complete atrial ventricular block (Cardiac disorders) | 14 (14) | 13 (13)
Asystole (Cardiac disorders) | 33 (33) | 41 (41)
Transfusion associated cardiac overload (Cardiac disorders) | 23 (23) | 8 (8)
Stroke (Nervous system disorders) | 26 (26) | 30 (30)
Transient ischemic attack (Nervous system disorders) | 3 (3) | 5 (5)
Pulmonary embolism or deep venous thrombosis (Vascular disorders) | 34 (34) | 26 (26)
Acute hemolytic transfusion reaction (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaphylactic transfusion reaction (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Pneumonia or Bacteremai (Infections and infestations) | 153 (153) | 166 (166)
Transfusion associated sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 153 (153) | 148 (148)
Acute renal failure (Renal and urinary disorders) | 233 (233) | 233 (233)
Transfusion related acute lung injury (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal Transfusion Strategy (N=1755) | Restrictive Transfusion Strategy (N=1749)
Atrial Fibrillation (Cardiac disorders) | 187 (187) | 194 (194)
Stable Angina (Cardiac disorders) | 183 (183) | 176 (186)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02981407/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02981407/SAP_002.pdf
  • Informed Consent Form (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT02981407/ICF_000.pdf